CLINICAL TRIAL: NCT03962192
Title: High-Intensity Specialist-Led Acute Care (HiSLAC) Project
Brief Title: Attitudinal Measures Survey With HISLAC Physicians (SURVEY ONLY)
Acronym: HiSLAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RG_13-251
Record Dates: First submitted 2019-05-03; First posted 2019-05-23 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2019-04

CONDITIONS: Attitude; Risk-Taking
MeSH Terms: conditions — Behavior; Risk-Taking

STUDY DESIGN:
Intervention Model Description: An attitudinal survey will be completed by approximately 80 case note reviewers within the HiSLAC project
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey tools (Experimental): Survey instruments are shared with reviewers.
  Interventions: Other: Attitudinal measures

INTERVENTIONS:
Other: Attitudinal measures — A collection of 3 distinct attitudinal instruments comprise this survey.

SUMMARY:
HiSLAC is an independent, professionally-led study which will evaluate a key component of NHS England's policy drive for 7-day services: the intensity of specialist-led care of emergency medical admissions, with a particular focus on weekend provision. This research is important for patients and for NHS strategy because it offers a unique opportunity to evaluate the impact of the transition to seven-day working, and to understand factors likely to impede or enhance the effectiveness of this change in practice.

In addition to examining the impact on patient-centred outcomes, the project will also undertake a health economics analysis of the impact of increasing specialist provision across the NHS. HiSLAC will therefore provide useful information across the NHS about the cost-effectiveness of investing in consultant and other specialist staffing in implementing the drive to 7-day service provision.

In this survey instrument, physician characteristics and psychological attitudes have been shown to influence medical decisions. This study aims to describe the influence of several patient characteristics and reviewer characteristics and attitudes on the physician's overall case note review care quality judgement using an analytical method called multi-level modelling.

DETAILED DESCRIPTION:
The investigators describe here a protocol for comparing quality of care given to patients admitted as emergencies to 20 hospital Trusts at weekends and on weekdays during two epochs, representing periods before (2012-2013) and during (2016-2017) the implementation of NHS England's 7-day services standards.

Using retrospective review of case records from 20 hospital Trusts during two time epochs, this study aims to determine whether there is a difference in quality of care offered to patients undergoing emergency admission (EA) to hospital at weekends compared with weekdays.

The main objectives are as follows:

1. To compare rates of errors and differences in care quality between weekend and weekday admissions,
2. To examine prevalent error types for weekend and weekday admissions,
3. If a difference in error rates or care quality between weekend and weekday admissions is found, examine whether the difference has changed between the two epochs.
4. To inform the Bayesian model proposed in this parallel health economics model. The co-primary outcomes are the weekend:weekday error rate ratio and the global assessment of care quality. The error rate is calculated as the number of errors per case record from admission to discharge or to 7 days, whichever occurs first.

Secondary outcomes include a comparison of weekend-weekday admissions in error typology and error-related adverse events (AEs), of error rates by day of the week within each admission group and correlation of weekend: weekday error rate ratios with weekend:weekday differences in specialist hours per 10 EAs.

In this survey instrument, physician characteristics and psychological attitudes have shown to influence medical decisions. The case note review process of determining the overall care quality is a type of medical decision. The HiSLAC study gives us an opportunity to determine whether patient or physician characteristics and physician attitudinal scores (physician aversion to ambiguity, need for cognition and personal need for structure) influence the overall care quality judgement during case note review. The investigators develop a case for considering this question with a multi-level model assuming the clustering within patient and within reviewers; furthermore, the investigators develop pre-specified hypotheses for testing. (See hypotheses) Our outputs from this are intended to inform better practice with case note reviews.

HYPOTHESES

For each objective a general hypothesis is provided:

Null hypothesis 1: To assess whether there is no significant relationship between patient case note characteristics and the physician's overall care quality judgements.

Null hypothesis 2: To assess whether there is no significant relationship between case note reviewer characteristics and their overall care quality judgements.

Null hypothesis 3. To assess whether there is no significant relationship between case note reviewer attitudes and their overall care quality judgements.

In addition to the above two objectives, one secondary objective is to assess the same effects of characteristics and attitudes on reviewer confidence in their care quality judgement. A further secondary objective is to assess whether there is a significant relationship between case-specific factors and reviewers' self-assessed confidence in their global care quality judgements.

ELIGIBILITY:
Inclusion Criteria:

* case note reviewer involved in the HiSLAC study (including those partly reviewing their apportioned cases.)

Exclusion Criteria:

* participants not involved at the outset or at any point during the HiSLAC case note reviews

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Need For Cognition (NFC) Scale (5 items on 6 point Likert) | 3 weeks from survey commencement
  Assessing the individual's tendency to engage in and enjoy activities that require thinking. Minimum score is 1 and the maximum is 6 (other than for items 3 and 4 which are each reverse scored; i.e. 6 is the lowest score and 1 is the highest score possible) There is no moral distinction about which score is better; they are measures of attitudinal predispositions individuals have in a respective scenario. It is then our remit to parse this information in light of the context, the nature of the participants and the overall aims and boundaries of reviewing case notes. (e.g. a higher value (thus preferring more complex situations) on 'I would prefer complex to simple problems' does not necessarily indicate a 'good' response but more that they are compelled by difficult and complex problems.
  There are no subscales to consider; items are equally weighted contributing to the distinction between low and high NFC i.e. top half or the bottom half of all possible scores.
Personal Need for Structure (PNS) Scale (12 items on 6 point Likert) | 3 weeks from survey commencement
  Assessing preferences for "structure and clarity in most situations, with ambiguity and grey areas proving troublesome and annoying." Minimum score is 1 and the maximum is 6 (other than for items 2, 5, 6 and 11 which are each reverse scored; i.e. 6 is the lowest score and 1 is the highest score possible) There is no moral distinction about which score is better; they are measures of attitudinal predispositions individuals have. Investigators then parse this information in light of the context, the nature of the participants and the overall aims and boundaries of reviewing case notes. (e.g. a higher value (thus preferring more complex situations) on 'I enjoy having a structured mode of life.' does not necessarily indicate a 'good' response but more that they desire more structure in their work.
  There are no subscales to consider for PNS; items are equally weighted contributing to the distinction between low and high PNS i.e. in the top half or the bottom half of all possible scores.
Anxiety due to uncertainty Scale (ADTU) (5 items on 6 point Likert) | 3 weeks from survey commencement
  One subscale (total=4) of 'Revised Physician's reactions to uncertainty scale' assessing physicians" affective reactions to uncertainty.
  Minimum score is 1 and the maximum is 6 (other than for items 2, 5, 6 and 11 which are each reverse scored; i.e. 6 is the lowest score and 1 is the highest score possible) There is no moral distinction about which score is better; they are measures of attitudinal predispositions individuals have. It is then our remit to parse this information in light of the case note review context. (e.g. a higher value (thus preferring more complex situations) on 'I am quite comfortable with the uncertainty in patient care' does not necessarily indicate a 'better' response but more that they are more comfortable with uncertainty in their clinical work.
  ADTU is a subscale of the a larger instrument; items are equally weighted contributing to the distinction between low and high ADTU i.e. in the top half or the bottom half of all possible scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Applied Health Research, University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The plan is to share the information once the data has been collected and cleaned. Researchers will be contacted to determine the next steps to be taken with the data. Analysis will occur and this will be shared with participants and researchers alike.

REFERENCES:
- See also: HiSLAC Study website — https://www.hislac.org/